#### **INFORMED CONSENT FORM**

THE PREVENT ANAL CANCER (PAC) SELF-SWAB STUDY

NCT Registration Number: NCT03489707

January 3, 2022-October 11, 2022

**Informed Consent for Research** 

Clinical Interventions template - Version: March 30, 2018

IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

# Medical College of Wisconsin and Froedtert Hospital INTRODUCTION TO THE INFORMED CONSENT

| Name of Participant: |
|----------------------|

Prevent Anal Cancer Study

Alan G. Nyitray, PhD
Department of Psychiatry and Behavioral Medicine
Center for AIDS Intervention Research & Clinical Cancer Center
414-805-3312
Medical College of Wisconsin
8701 Watertown Plank Road
Milwaukee WI 53226

You are invited to take part in this research. You can decide whether to take part in this project or not. You are free to say yes or no. If there is anything that you do not understand, please ask questions.

#### **Definitions**

Anal canal – the part of the body that starts at the opening of the anus and goes into the body for 1-2 inches.

DARE – during a digital anal rectal exam the doctor/nurse views the perianal region and inserts a finger into your anus to look and feel for disease.

Human papillomavirus (HPV) – a virus that causes most anal cancers.

High-resolution Anoscopy (HRA) – a medical procedure where a health care provider (HCP) inserts a scope into the anus to see if there are changes that can lead to cancer.

Methylation – a process by which molecules are added to DNA. It is not known at this time if methylation will help identify persons at increased risk for anal cancer.

Cis-man – a person who identifies as a man and was assigned a male sex at birth.

**Informed Consent for Research** 


IRB Protocol Number: <u>00032999</u>

IRB Approval Period: 1/3/2022 - 10/11/2022

#### **EFFECTIVE**

1/3/2022

MCW/FH IRB

#### **Purpose**

This project is being done to learn about ways to test for anal cancer in gay and bisexual cismen and transgender persons.

#### Length

You will be in this research project for 3 visits over about one year. The total time commitment during the year is 2.5 – 3 hours.

If it was found that you should have treatment, we would also like to keep in contact until you finish your treatment.

#### **Procedures**

We will first give you a survey and then put you in one of two groups.

- People in group one are mailed an anal self-swabbing kit to use at home. After using the kit, they'll mail it back to us, take a survey, and then go to a HCP who will measure weight, height and waist circumference andprovide a digital anal rectal exam (DARE) and an anal swab. Then they'll take a survey.
- 2) People in group two will go to a study clinic where a HCP will measure weight, height and waist circumference and provide a digital anal rectal exam (DARE) and and an anal swab. Then they'll take a survey.

Swabs from both groups will be sent to a lab for testing.

One year later, people in both groups will do the same procedures again. Then, they will have high-resolution anoscopy (HRA) with biopsies along with one final survey.

#### List of visits:

- Virtual Consenting and online baseline survey
- -Total Number: 1
  - -Total time: 30 min
  - Visit 1
    - -Total Number: 1
    - -Time:Group 1-15 min; Group 2-20 min
- Visit 2-Total Number: 1
- -Time: Group 1(no visit); Group 2-20 min

#### Risks

This is a brief list of the most common potential research risks. The *full consent form* after this introduction contains a more complete list of potential research risks.

#### Intervention risks:

Embarrassment answering questions on a survey.

Discomfort and/or embarrassment during

- anal canal swabbing
- DARE
- HRA

Irritation and/or some bleeding during biopsies.

Disclosure of confidential information.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

Visit 3 - HRA

-Total Number: 1

-Total Time: Both Groups-20 min

# Procedures that will occur at various visits:

#### **Invasive Procedures**

- Visit 1-anal swab and DARE
- Visit 2-anal swab and DARE
  - -Total Number: 1
  - -Time: Group 1-no visit; Group 2- 25 min
- Visit 3-HRA with a minimum of 2 biopsies

#### **Non-invasive Procedures**

Surveys

This project may or may not help you, but we hope the information from this project will help us develop a better screening process for anal cancer.

### **My Other Options**

You do not have to join this project. You are free to say yes or no.

- Whether or not you join this project, you are free to seek services from this or other agencies.
- Whether or not you join this project, your usual medical services will not change.

If you have more questions about this project at any time, you can call Alan G. Nyitray, PhD at 414-805-3312.

If you have questions about your rights as a participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

#### CONSENT TO PARTICIPATE IN RESEARCH

#### A1. INTRODUCTION - WHY ARE WE ASKING YOU TO PARTICIPATE?

You are being invited to participate in this research because you are a resident of the Milwaukee metro area, identify your gender as either male or transgender person and are aged 25 years or older. To be eligible, you also must acknowledge sex with cis-men in the last five years <u>or</u> identify as gay or bisexual.

Persons who are not eligible for the study:

- Persons with a prior diagnosis of anal cancer
- Persons who use anticoagulants or blood thinners
- Persons not willing to attend one of the Milwaukee study clinics
- Persons who plan to move in the next 12 months

A total of about 500 persons in Milwaukee are expected to participate in this research.

The Director of the project is Alan G. Nyitray, PhD in the Medical College of Wisconsin Cancer Center and the Center for AIDS Intervention Research. A research team works with Dr. Nyitray. You can ask who these people are.

The National Institutes of Health, a government agency, is funding the research.

#### **A2. DO I HAVE TO PARTICIPATE?**

You can decide whether to take part in this research or not. You are free to say yes or no. If you say no, your regular medical care will not change. Even if you join this project, you do not have to stay in it. You may stop at any time.

A research project is different from routine medical care in two ways: 1) there are extra risks that we will tell you about in this form; 2) the research procedures, tests and visits follow a set plan that must be kept.

#### A3. WHY IS THIS PROJECT BEING DONE?

In this study, we want to learn about the best ways to create screening programs for anal cancer. Anal cancer screening is not widely recommended for public health programs. But if screening is going to be recommended in the future, 1) we want to learn what might be a better way to do public health screening and 2) we want to learn more about tests that could help identify people at increased risk for anal cancer.

To learn about a better way to do screening, we want to know if persons prefer screening at home or screening at a doctor's office. Half of the persons in this study will be asked to do screening at home by self-swabbing the anal canal, and the other half will be asked to get the swabbing done by a Health Care Provider (HCP) at a clinic.

To learn about tests that may help identify who is at increased risk for anal cancer, the swabs will be tested for HPV persistence and for methylation. Both of these are experimental, and neither is approved by the U.S. Food and Drug Administration (FDA) for use in the clinic.

#### **Informed Consent for Research**


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

#### **EFFECTIVE**

1/3/2022

MCW/FH IRB

Neither is routinely used in clinics to help screen for anal cancer because it's not known if they will help.

Finally, public health screening programs may include DARE and HRA. We want to know what you think about these procedures.

#### **B1. WHAT WILL HAPPEN IF I PARTICIPATE?**

If you decide to be a part of this research, during this remote consenting session we'll collect your address and other contact information. Then we'll ask you to fill out a baseline survey (15 mins – also online) that will ask you questions about anal cancer screening, sexually transmitted infections, and sexual behavior. If you complete this survey, we will enroll you in the study and ask for your contact information so we can send you study materials.

The following are activites that everyone in the study will do:

- We will measure everyone's height, weight and waist circumference
- Persons who are HIV-negative or HIV-unknown will get an HIV test at the beginning of the study and one year later.
- Everyone will complete surveys after anal canal swabbings (5 minutes), and after HRA (5 minutes).

#### Research groups

Because no one knows which of the screening interventions is best, you will be randomized into one of two groups. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance of being placed in either group. Neither you nor the research investigator can choose what group you will be in. We'll notify you which group you are in after you've completed the baseline survey.

1) For people in group one, we will mail a self-swabbing kit to your home within 2 weeks of enrollment. This kit was designed by the study because no commercial kit for anal self-swabbing for gay and bisexual men and trans persons exists. When you receive the kit, you will read the instructions and then use a swab (like a large Q-tip) to swab your anal canal. Reading the instructions and using the swab will take 5 - 10 mins. The swab will go into the anal canal about 3 inches. You will then send the swab back to us. Then, we'll ask you to go to a HCP at one of five Milwaukee clinics for a DARE and another anal canal swab (10 mins). If the HCP is concerned about anything when doing the DARE, the HCP will tell you and provide referrals to care, if needed.

The study clinics are

Vivent Health (formerly AIDS Resource Center of Wisconsin), Milwaukee, WI Anal Dysplasia Program of MCW-Froedtert, Milwaukee, WI Holton Street Clinic, Milwaukee, WI Inclusion Clinic of MCW-Froedtert, Milwaukee, WI Sixteenth Street Community Health Centers, Milwaukee, WI

#### **Informed Consent for Research**


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

#### **EFFECTIVE**

1/3/2022

MCW/FH IRB

2) For people in <u>group two,</u> we will ask you to go to one of the five study clinics above within 2 weeks of enrollment. There, a HCP will swab your anal canal and do a DARE just like group 1. The swabbing and DARE will take about 10 mins.

At the end of the visits for both group one and group two, we'll tell you about the study's voluntary referral program which provides incentives for referring your friends and family to the study.

We will send swabs from both groups for testing that is experimental: testing for human papillomavirus (HPV) DNA and host/virus methylation. These two tests have no clinical value at this time. In other words, the results of a single test are not known to be useful in determining risk for anal cancer.

One year later, we will ask you to do the same procedures again: persons in group one will get a swabbing kit in the mail (we'll let you know when it's about to be mailed); persons in group two will be asked to go to a clinic for a swabbing. Persons in each group will again tell us about their experiences doing the screening.

Then, all persons will have high-resolution anoscopy (HRA) and DARE which will be done at the MCW-Froedtert Anal Dysplasia Program which will also help you know if you are at increased risk for anal cancer. This will take about 15 mins. HRA is the gold standard for detecting problems in the anal canal that could put a person at risk for anal cancer. HRA involves inserting an anoscope into the anus so that the HCP can assess the health of your anal canal. The procedure includes putting a weak vinegar solution on the anal canal walls to help the HCP see if there are any problems. If the HCP can't see any problems in your anal canal, the provider will take two biopsies so that they can be examined further by a specialist doctor in detecting cancer to better establish that there are no problems. If there are areas of concern in your anal canal or perianal tissue, the HCP will biopsy those areas of concern so that they can be examined further by the specialist. The HCP will give you the results of the HRA and tell you if there is a need for follow up. You'll also complete a final survey about your HRA experience which takes about 5 mins. When the biopsies have been examined, we'll give you those results too.

We will do a blood draw during the HRA visit. The blood specimen will allow us to test for factors in your blood, like HIV, that are, or may be, associated with anal precancers. If the HIV test is positive, we will inform you, and report your HIV status to government health agencies as required by law. Results of your blood test will be used in this study to better understand factors associated with anal precancers and released only to authorized persons as governed by Wisconsin law. HIV test results of active military personnel will be forwarded to the military medical authority of the base to which you are assigned, as required by the Department of Defense.

As mentioned above, the swabbing that you or the HCP will do includes checking for human papillomavirus (HPV). HPV in the anal canal is very, very common but only a very small percentage of persons with anal HPV are at risk for anal cancer. Since a one-time HPV test is not FDA-approved, is probably not helpful for knowing the risk for anal cancer, and takes at least six months for results, we will not be able to give you the first anal canal swabbing results. You will be given results if there is evidence of 12-month high-risk persistence, that is if you

#### **Informed Consent for Research**


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

#### **EFFECTIVE**

1/3/2022

MCW/FH IRB

have had the same high-risk HPV type during the past year. These results will not be available until 3-9 months after your HRA. Results of the methylation test will not be given to you since it is experimental and not known to be useful in assessing risk for anal cancer.

#### **Summary of Procedures:**

Here's what to expect as a participant if you agree and are able to take part in this study:

- 1) You will complete a survey online (or on paper if you have no Internet access).
- 2) You will be placed into a group that will get a kit in the mail for anal canal swabbing or a group that will be asked to go to a clinic for anal canal swabbing.
- 3) Persons in both groups will get a DARE and anal swabbing at a clinic.
- 4) Persons in both groups will complete surveys about their experience with swabbing and DARE.
- 5) Persons in both groups will do the swabbing and DARE again in one year and tell us about the experience in a survey.
- 6) Persons in both groups will get HRA which is the gold standard for knowing if a person is currently at risk for anal cancer. We will tell you the results. You will tell us about the HRA experience in a survey.
- 7) If you have high-risk HPV persistence, as confirmed by the swabbing over one year, we will give you these results within nine months after the HRA.

#### **B2. HOW LONG WILL I BE IN THE PROJECT?**

You will be in this research project for about 1 year. The total amount of time you will take part in this research study during the year is about 2.5 to 3 hours.

After the study is finished, we want to keep in touch with you to follow your health over time. We will telephone you once a year for two years and ask about screening for anal cancer that you may have done on your own and the results of that screening.

#### **B3. CAN I STOP BEING IN THE PROJECT?**

You are free to withdraw from the project at any time. If you leave, your regular medical care will not change. If you are thinking about leaving, please tell the research investigator.

The research investigator may take you out of this project at any time. This would happen if:

- They think it is in your best interest.
- You do not follow the project rules.
- The whole project is stopped.

If this happens, the research investigator will tell you.

#### **B4. ARE THERE ANY SPECIAL INSTRUCTIONS WHILE I AM IN THE PROJECT?**

If you begin to take prescription blood thinners or anti-coagulants during the study, it is important to let the research investigator know before you get the HRA. We also ask you to not

#### **Informed Consent for Research**


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

#### **EFFECTIVE**

1/3/2022

MCW/FH IRB

have receptive anal sex in the 24 hours before getting an anal swabbing, either a self-swabbing or a clinician swabbing.

#### C1. WHAT HEALTH RISKS OR PROBLEMS CAN I EXPECT FROM THE PROJECT?

We watch everyone in the project for problems (side effects). You need to tell the research investigator or a member of the research team immediately if you experience any problems. If you have severe bleeding after the HRA, call Advance Practice Nurse Practitioner Sarah Lundeen immediately at 414-955-5783. In an emergency, call 911.

The possible risks to you in this study can be divided into four groups: a) risks during the swabbing, b) risks during the DARE, c) risks during HRA, and d) discomfort with sensitive questions.

- a) <u>The swabbing.</u> The insertion and rotation of the swab (like a Q-tip) may be slightly uncomfortable.
- b) The HCP will give you a DARE in the study. This means the HCP will look at your perianus for signs of disease. Then the doctor/nurse will put lube on their index finger, and then insert the gloved finger into your anal canal. The doctor/nurse will put a finger approximately 2-3 inches inside of you and feel for something that is not normal. While this is a common and safe procedure often used in physical exams, it may be mildly uncomfortable or embarrassing to some people.
- c) <u>HRA.</u> The procedure of inserting the scope into the anal canal may be embarrassing for some persons. The anal speculum can be uncomfortable, and the vinegar solution can cause some irritation in the anus. Some bleeding occurs with every biopsy. Serious bleeding is rare, about 1 in 1000 biopsies. If serious bleeding occurs, a simple procedure may be necessary to stop the bleeding such as burning or cauterizing the area. An injection of lidocaine may be given prior to a biopsy. It is possible to experience pain or dizziness from the injection. Rarely, an allergic reaction could occur.
- d) <u>Discomfort with sensitive questions.</u> This study will ask survey questions about sexual behavior, disease status and alcohol and drug use. Some people may feel embarrassed in answering these questions on the survey. You may get tired when you are completing a survey; however, you do not have to answer any questions you do not want to answer.

Another risk may be loss of confidentiality. Every effort will be made to keep your research records confidential but we cannot guarantee it. Depending on the kind of information being collected, if your research information were accidentally seen, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the project director about whether this could apply to you.

So it is possible that someone could find out that you were in the study and learn something about you that you did not want them to know. But this is very unlikely because we will do everything we can to keep your information private.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

#### C2. OTHER RISKS OF THIS RESEARCH PROJECT

Screening for anal cancer is not yet recommended because it may do more harm than good. For example, it's possible that you may have a biopsy that indicates there is a risk for anal cancer when there really is no risk. This could cause unnecessary anxiety and medical tests.

#### C3. ARE THERE ANY BENEFITS TO TAKING PART IN THE PROJECT?

At the beginning of the study and at the end of the study, a highly-experienced HCP will examine you for signs of anal cancer. This may help you learn of an anal condition or disease for which you need treatment. If any problems are found, the HCP will give you the results and recommend places for follow up and/or treatment.

Your participation in this study may help us learn more about the most effective ways to do anal cancer screening.

#### D1. ARE THERE ANY COSTS TO BEING IN THE PROJECT?

There are no costs to you for the <u>study activities</u> you do as part of this study. They are free. The study activities that are paid for by this study are anal swabbing, DARE, HRA, and biopsies done during the HRA. In addition, the study will pay for a specialist doctor to review the biopsies to determine if there is any disease present. You will also not have to pay for tests done on the swab. If you have questions regarding costs, please contact Dr. Alan Nyitray.

It's possible that at a study visit you may be offered services that are not part of this study. For example, the study HCP could find something after doing your DARE and recommend treatment and follow-up care. That treatment and follow-up care will not be reimbursed by this study; however, those costs can be billed to a third-party payer like your insurance, Medicare, or Ryan White.

If you receive a bill that you believe is related to your taking part in this research study, please contact Dr. Alan G. Nyitray 414-805-3312 with any questions. Do not pay the bill.

If you participate in this research, the costs of any necessary emergency medical treatment in the event of a research-related injury will be billed to you or your health insurance.

#### D2. WILL I BE PAID FOR PARTICIPATING IN THE PROJECT?

You will be compensated as follows for various parts of the study:

\$35 at the baseline swab and survey.

\$45 at the 12-month swab and survey.

\$50 at the HRA and survey.

Therefore, if you complete the entire study, you would be compensated for a total of \$130. Any payment may be reportable as income on your taxes.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

#### D3. WHAT OTHER HEALTHCARE CHOICES DO I HAVE?

You do not have to join this project. You are free to say yes or no. If you do not join this project, your research investigator can discuss other healthcare choices with you.

You may be able to get some of the procedures used in this research through other HCPs.

The research investigator can explain both the possible benefits and the risks of other options that are available to you.

#### D4. WILL I BE GIVEN NEW INFORMATION ABOUT THE PROJECT?

If we learn any important new information about anal cancer screening that might change your mind about being in the project, we will tell you about it right away. You can then decide if you want to stay in the project.

Clinically relevant results, including individual results, for DARE, HRA, and HPV persistence, will be disclosed to you. The HCP who does the DARE and HRA will tell you if there is anything that is found that should be followed up. The study staff will tell you after the HRA if there was high-risk persistence for HPV. But persistence is very common and most people who have persistence will never get anal cancer.

#### D5. WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THE PROJECT?

Emergency medical treatment for injuries directly related to your participation in this research project will be provided to you. You or your health insurance will be billed for the costs of this emergency treatment. MCW will decide on a case by case basis if they will reimburse you or your insurer for emergency treatment costs. If your research-related injury requires medical care beyond this emergency treatment, you or your insurer will be responsible for the costs of this follow-up care.

At this time, there is no plan for any additional financial payments.

If you believe that you have been injured because of your participation in this project, contact the research investigators right away. Contact information: Principal Investigator Dr. Alan Nyitray at 414-805-3312.

Nothing in this consent form affects any legal rights you may have nor does it release the investigator, the sponsor, the institution, or its agents from liability for negligence.

#### D6. WHO CAN ANSWER MY QUESTIONS ABOUT THE PROJECT?

- If you have more questions about this project at any time, you can call Principal Investigator Dr. Alan Nyitray at 414-805-3312.
- If you have questions about your rights as a research participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

# E. PERMISSION TO COLLECT, USE AND SHARE HEALTH INFORMATION E1. What health information will be collected and used for this project?

To be in this research project, the research team needs your permission to access, collect and use some of your health information. If you say no, you cannot be in the project. This information may come from questions we ask, forms we ask you to fill out, or your medical record, as described below. We will only collect and use information needed for the project.

The protected health information (PHI) originates from services you will or have received at one or more of the following locations: the Medical College of Wisconsin (MCW); BloodCenter of Wisconsin (BCW); Children's Hospital of Wisconsin (CHW); any Froedtert Health Affiliate-Froedtert Memorial Lutheran Hospital (FMLH), Inc.; Community Memorial Hospital (CMH) Menomonee Falls, Inc.; St. Joseph's Community Hospital (SJH) West Bend, Inc.; Froedtert & The Medical College of Wisconsin Community Physicians Clinics, Inc. (FMCWCP); the West Bend Surgery Center, LLC; and the Froedtert Surgery Center, LLC.

### The health information to be collected and used for this project is:

Health status. For example, we will ask if you have ever had anal cancer or if you are HIV-positive.

Information on medical records of the care you receive for this project.

Information on prior medical records about anal cancer screening or HPV-associated disease.

Information on medical records dating from when you join this project until two years after its conclusion.

#### E2. Who will see the health information collected for this project?

The only MCW/Froedtert Hospital employees allowed to handle your health information are those on the research team, those on the Institutional Review Board (IRB) and those who check on the research activities to make sure the hospital's rules are followed.

If the costs of any necessary emergency medical treatment in the event of a research-related injury are billed to your health insurance, your health information may need to be disclosed to the insurer for billing purposes.

The research team may share your information with people who don't work at MCW/Froedtert Hospital because they planned, pay for, or work with us on this project. The federal Privacy Rule may no longer protect your health information once it leaves MCW/Froedtert Hospital. For this project, we plan to share information with those doctors, researchers or government representatives working with us on this project at the institutions or companies listed here:

In this study, you will choose to get clinical services at one of the following Milwaukee clinics. The results of DARE, HRA and results of persistence testing for high-risk HPV will be provided to the clinic that you decide to go to for clinical services as part of this study.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

Vivent Health, Milwaukee, WI Anal Dysplasia Program of MCW-Froedtert, Milwaukee, WI Holton Street Clinic, Milwaukee, WI Inclusion Clinic, Milwaukee, WI Sixteenth Street Community Health Center, Milwaukee, WI

MCW is a medical school. Once all personal identification is removed from your biopsies, we may use images of your biopsies to train medical students, residents and fellows on how to recognize tissue changes that may lead to anal cancer.

We may record your research information, including results of tests and procedures done for research, in your Froedtert Hospital and/or Medical College of Wisconsin medical record. As a result, this research information may be seen by people allowed to see your medical records for healthcare operations or treatment, by those you allow to see your medical records by giving written permission, and by others when required by law.

We will not use your personal health information for a different project without your permission or the permission of a hospital research review board (IRB). Once all personal identification is removed from your health information and/or biospecimens, the information and/or biospecimens may be used for future research or distributed to another investigator for future research without additional informed consent from you or your legally authorized representative. The information might also be used or released for other purposes without asking you. Results of the project may be presented in public talks or written articles, but no information will be presented that identifies you.

#### **E2.5 Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The study team can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena.

The study team will use the Certificate to resist any demands for information that would identify you, except the following:

The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

#### E3. What are the risks of sharing this health information?

One risk of taking part in a research project is that more people will handle your personal health information collected for this project. This means it is possible that someone could find out that

Medical College of Wisconsin & Froedtert Hospital **Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

you were in the study and learn something about you that you did not want them to know. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the research investigator about whether this could apply to you.

#### E4. How long will you keep the health information for this project?

If you sign this form, we plan to keep your information for 10 years after the research project ends in case we need to check it again for this project.

#### E5. Can I cancel my permission to share this health information?

If you change your mind later and do not want us to collect or share your health information, you need to send a letter to Dr. Alan Nyitray at the Medical College of Wisconsin, *Clinical Cancer Center, Suite 5400, 8701 Watertown Plank Road, Milwaukee, WI 53226-3548.* The letter must say that you have changed your mind and do not want the researcher to collect and share your health information. At that time, we may decide that you cannot continue to be part of the project. We may still use the information we have already collected.

#### F1. FOR MORE INFORMATION ABOUT THE PROJECT

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can look up this project by referring to the ClinicalTrials.gov number (NCT03489707) or by asking the research team for a printed copy.

**Informed Consent for Research** 


IRB Protocol Number: 00032999

IRB Approval Period: 1/3/2022 - 10/11/2022

**EFFECTIVE** 

1/3/2022

MCW/FH IRB

#### **CONSENT TO PARTICIPATE**

#### By signing my name below, I confirm the following:

- I have read (or had read to me) this entire consent document. All of my questions have been answered to my satisfaction.
- The project's purpose, procedures, risks and possible benefits have been explained to me.
- I agree to let the research team use and share the health information and other information gathered for this project.
- I voluntarily agree to participate in this research project. I agree to follow the procedures as directed. I have been told that I can stop at any time.

**IMPORTANT:** You will receive a signed and dated copy of this consent form. Please keep it where you can find it easily. It will help you remember what we discussed today.

| Subject's Name please print | Subject's Signature | Date |
|-----------------------------|---------------------|------|